CLINICAL TRIAL: NCT06143124
Title: Bismuth Quadruple Therapy Versus Standard Triple Therapy for the First-line Treatment of Helicobacter Pylori Infection in Children: Efficacy and Safety
Brief Title: Bismuth Quadruple Therapy Versus Standard Triple Therapy
Acronym: BismoHelP
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Tadej Battelino, Clinical Professor, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BismoHelP
Record Dates: First submitted 2023-11-04; First posted 2023-11-22 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Helicobacter Pylori Infection
Keywords: children; eradication therapy; antibiotics
MeSH Terms: interventions — bismuth tripotassium dicitrate

STUDY DESIGN:
Intervention Model Description: one group (control) the classical eradication treatment therapy (14 days), second group (therapeutic) shorter duration of therapy (7 days) with the same drugs including Bismuth
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapeutic arm (Active Comparator): Classical triple therapy according to the antibiotic susceptibility testing (two antibiotics+PPI)+ Bismuth subcitrate for 7 days
  Interventions: Drug: Bismuth Subcitrate
- Control arm (No Intervention): Classical triple therapy according to the antibiotic susceptibility testing (two antibiotics+PPI) for 14 days

INTERVENTIONS:
Drug: Bismuth Subcitrate — shorter duration of therapy (7 instead of classical 14 days) with four dugs instead of three (adding Bismuth subcitrate).
  Arms: Therapeutic arm

SUMMARY:
The goal of this clinical trial is to compare the standard triple therapy with Bismuth quadruple therapy in children infected with Helicobacter pylori.

The main questions to answer are:

* the safety
* the efficacy of the quadruple protocol with Bismuth subcitrate

Participants will be randomised in 7-days eradication therapy group and 14-days eradication control group.

DETAILED DESCRIPTION:
Infection with Helicobacter pylori (H. pylori) is still a very common bacterial infection in humans, despite the worldwide significant decrease in incidence and prevalence recorded in recent years. Infection with H. pylori is mostly acquired during early childhood, and in low prevalence countries such as European countries, infected family members, particularly the mothers, are the main source of infection. Chronic inflammation of the gastric mucosa can cause peptic erosions and ulcerations, gastric adenocarcinoma and mucosa-associated lymphoid tissue lymphoma. In addition, extra gastric complications, such as iron-deficiency anemia, may be induced by H. pylori infection. The first line treatments currently available for children infected with H. pylori are various combinations of proton pump inhibitors (PPI) with antibiotics including amoxicillin, clarithromycin and/or imidazoles. While previously 7 days treatment had been recommended, the low eradication rate demanded longer treatment duration of 10-14 days increasing the chance for adverse effects and lower compliance to therapy.

In the last decade, the eradication rates using these schemes have declined and have led to recommendation for higher dosages, longer duration of therapy or regimens including three instead of two different antibiotics, either sequentially or concomitantly. The low success rates are essentially due to the increasing resistance rates to macrolides and to lesser extent imidazole. Koletzko et al. detected very high primary resistance rates to metronidazole and clarithromycin in Europe (23% and 20%, respectively), whereas resistance after failed eradication therapy was even higher (35% and 42%, respectively). Children born to mothers from developing countries and Asia have extremely high primary resistance rates to metronidazole due to the frequent usage of this drug for parasitic infection in Africa and Asia. The high resistance rate to clarithromycin is caused by the frequent use of macrolides in children for respiratory tract infections resulting in a higher primary clarithromycin resistance rates in paediatric patients compared to adults. The newest guidelines of the European and North American societies of Gastroenterology, Hepatology and Nutrition (ESPGHAN and NASPGHAN) recommend in anti - H. pylori infected children to perform culture and antibiotic susceptibility testing prior first therapy and to tailor the therapy according to the results, and give higher doses as previously suggested with a treatment duration of 14 days.

Adverse events such as diarrhoea, nausea, taste disturbance, and abdominal pain are frequent during eradication therapy and mainly due to antibiotics, with diarrhoea being the most common one. Higher doses and longer treatment duration recommended in the newest guidelines may augment this problem and may result in discontinuation of the therapy. Since non- compliance to therapy is the second most frequent cause for treatment failure improving compliance by decreasing adverse effects may result in better clearance rates with a lower risk for the development of antibiotic-resistance strains.

Therefore, new therapeutic protocols are needed to decrease side effects and improve compliance for H. pylori treatment protocols and hopefully to raise the eradication rates.

The Bismuth salicylate is an option as part of first line therapy in children for H. pylori eradication already at the two latest paediatric guidelines NASPGHAN/ESPGHAN published in 2011 and 2017. BS is not used more in praxis due to the fact that is not available in the drugstores in many European countries. In Slovenia is it on the market in the form of Bizmut oksid 120 mg produced by Krka pharmaceutical company. It is officially registered for H. pylori eradication. There is a lot of data in adults, but very little prospective data in children available on the treatment protocols with BS and eradication rates in an anti-H. pylori therapy in a paediatric population. It is an investigator initiated single center, randomized, study to compare the effectiveness of triple therapy (PPI, two antibiotics (tailored to antibiotic susceptibility testing)) given for 2 weeks with the same eradication protocol (PPI, two antibiotics (tailored to antibiotic susceptibility testing)) lasting only for one week with Bismuth subcitrate in H. pylori infected children. The study included a pre-screening, an intervention (1-2 weeks) and a post-intervention time (8 weeks), with total of 2 visits and 2 phone calls after inclusion. The total duration of the study will be 8 weeks.

Subjects: Children aged 5 (>15 kg) -18 years, diagnosed with H. pylori infection during upper endoscopy with a positive culture and results for antibiotic susceptibility testing for clarithromycin and metronidazole and without resistance to both antibiotics who meet all inclusion and none of the exclusion criteria.

Symptoms (abdominal pain, bloating, nausea, vomiting, bad metallic taste) on the diary are scored from 0-3 (0=none; 1=mild, not interfering with normal activity; 2=moderate, interfering with normal activity; 3=severe, daily activity not possible). Stool pattern are monitored for frequency and consistency (0=no stool, 1=hard (Bristol stool scale 1-2), 2=formed (BSS 3-4), 3=soft (BSS 5-6), 4=watery (BSS 7). A number for each stool must be filled. We defined diarrhoea as more than two soft stools (Bristol stool scale 5 or 6) per day and/or one or more stools of watery consistency (BSS 7), and constipation as less than 3 bowel movements per week and/or stools of hard consistency. The intake drugs of the triple therapy, the study product and concomitant drugs are recorded on the diary. In addition, special events of interest will be recorded.

Randomization will be performed in two groups with sealed envelopes: group with 7-day therapy plus BS and group of patients with 14-days therapy without BS. The therapy will otherwise be prescribed according to the antibiotic susceptibility testing. Patients susceptible for clarithromycin will receive amoxicillin and clarithromycin, if resistant to clarithromycin they will receive amoxicillin and metronidazole. Double-resistant patients (not susceptible to neither Clarithromycin nor to Metronidazole) are excluded as mentioned above.

Once allocated, the children randomization numbers will be used to identify the participant during the study period. A child who, for whatever reason, withdraws or is withdrawn from the study after having been allocated a randomization number (R-code), will be classified as drop out and identified as such in the relevant report.

The patient will record the intake of study product and triple therapy in a diary on a daily basis. The adherence to the prescribed treatment will be checked at visit 2 and expressed in percent of doses taken. An adherence of >80 % will be considered as per protocol, an adherence <80 % is considered as protocol violation and these patients will be considered for ITT analysis.

ELIGIBILITY:
Inclusion Criteria:

* • Male or female patients

  * Age between 5 - 18 years with a
  * Minimum body weight of 15 kg
  * Endoscopy performed with biopsies taken for culture, histology
  * No previous therapy for H. pylori infection
  * Written informed consent
  * H. pylori infection confirmed by positive culture and with susceptibility testing for clarithromycin and metronidazole to allow tailored therapy

Exclusion Criteria:

* Significant acute or chronic gastrointestinal disease (IBD, coeliac disease, GERD etc.) or other organic disease interfering with symptom assessment

  * Patients with ulcers and need to be treated with PPI according to the physician judgment.
  * Known allergies to used antibiotics, proton pump inhibitors or probiotics
  * Having received treatment with antibiotics or bismuth compounds during the previous 30 days before endoscopy.
  * Having received proton pump inhibitors during the previous two weeks.
  * Severe acquired or primary immunodeficiency disorder
  * Language barriers which do not allow to give informed consent and/or to adequately complete the study diary
  * Being infected with a strain resistant to clarithromycin and metronidazole (double resistant)

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 216 (Estimated)
Dates: Start 2022-03-03 (Actual); Primary Completion 2025-11-03 (Estimated); Study Completion 2025-11-03 (Estimated)

PRIMARY OUTCOMES:
Adverse effects of the Bismuth | duration of treatment (7 days)
  questionnaire for possible side effects

SECONDARY OUTCOMES:
Eradication therapy success of 7 days treatment protocol | one months
  eradication therapy succes checked with stool antigen test at least one months after the treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Matjaž Homan, Ljubljana, Slovenia

REFERENCES:
- [Result] Homan M, Hojsak I, Kolacek S. Helicobacter pylori in pediatrics. Helicobacter. 2012 Sep;17 Suppl 1:43-8. doi: 10.1111/j.1523-5378.2012.00982.x. PMID 22958155
- [Result] Jones NL, Koletzko S, Goodman K, Bontems P, Cadranel S, Casswall T, Czinn S, Gold BD, Guarner J, Elitsur Y, Homan M, Kalach N, Kori M, Madrazo A, Megraud F, Papadopoulou A, Rowland M; ESPGHAN, NASPGHAN. Joint ESPGHAN/NASPGHAN Guidelines for the Management of Helicobacter pylori in Children and Adolescents (Update 2016). J Pediatr Gastroenterol Nutr. 2017 Jun;64(6):991-1003. doi: 10.1097/MPG.0000000000001594. PMID 28541262
- [Result] Butenko T, Jeverica S, Orel R, Homan M. Antibacterial resistance and the success of tailored triple therapy in Helicobacter pylori strains isolated from Slovenian children. Helicobacter. 2017 Oct;22(5):e12400. doi: 10.1111/hel.12400. Epub 2017 Jun 27. PMID 28653787